CLINICAL TRIAL: NCT06535724
Title: Endoscopic Debridement of Chronic Plantar Fasciitis With Heel Spur Resection: a Novel Technique With Promising Outcomes - a Prospective Cohort Study
Brief Title: Endoscopic Debridement of Chronic Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehasport Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSC_TPION_2024_V1
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Fasciitis, Plantar; Fasciitis, Plantar, Chronic; Heel Spur
MeSH Terms: conditions — Fasciitis, Plantar; Heel Spur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients underwent endoscopic debridement coupled with heel spur resection. This method emphasizes the removal of pathologically altered tissue while preserving the plantar aponeurosis, with the aim of minimizing procedural morbidity and enhancing recovery outcomes. It specifically targets the crucial roles of the plantar fascia in supporting the foot arch and facilitating foot propulsion. All had experienced persistent plantar fasciitis symptoms for at least six months despite conservative treatment.
  Interventions: Procedure: Chronic plantar fasciitis endoscopic debridement coupled with heel spur resection

INTERVENTIONS:
Procedure: Chronic plantar fasciitis endoscopic debridement coupled with heel spur resection — 1. Preoperative Preparation: popliteal nerve block, patient positioning supine with the operated limb fully externally rotated, spinal anesthesia, tourniquet application.
  2. Surgical Procedure:
     * Initial Marking from the heel bone arch to the calcaneal bone to locate the entry point.
     * First Incision and Portal Creation: an initial incision at the palpated site using a size 11 blade; blunt dissection to reveal the plantar fascia; arthroscope entry.
     * Secondary Entry: 3 cm distally from the initial incision; positioning of the arthroscope; additional blunt dissection and obturator insertion.
     * Operative Technique: continuous irrigation with sterile saline; 3.5-mm shaver introduced through the distal portal; meticulous debridement of inflamed and pathological tissue; removal of calcaneal spurs; thinning of the plantar fascia
  3. Postoperative Care • Careful monitoring and guided rehabilitation to support optimal healing and recovery.

SUMMARY:
The aim of the study was to prospectively evaluate the results of endoscopic treatment of chronic plantar fasciitis with resection of the heel spur. Treatment was assessed based on the results of clinical examinations and functional assessment as well as X-ray examination.

DETAILED DESCRIPTION:
Hypothesis: Conducting research on a group of patients will prove that the use of endoscopic technique with heel spur resection for the treatment of chronic plantar fasciitis will improve the functional results of the foot.

Methods: Patients diagnosed with chronic plantar fasciitis will undergo surgical treatment. An inspection is planned before and after 3, 6, 12, 24 and 60 months. During the check-up, the patient will undergo an X-ray examination, medical and physiotherapeutic assessment.

Study plan:

Participation in the research involves arriving at the Rehasport Clinic in Poznań on the dates set by the Chief Investigator (3, 6, 12, 24 and 60 months after the surgical treatment). During the visit, members of the research team ask participants to complete a set of questionnaires, perform a medical examination with a physiotherapeutic assessment described in detail below, and an X-ray examination. The entire examination will last approximately 3 hours.

1. During all visits to Rehasport Clinic, the participant will be asked to complete the surveys ACFAS ankle and foot assessment scale.
2. During the same visits, research team members perform the following tests and examinations:

   1. medical examination - aimed at assessing current ailments and range of motion,
   2. X-ray examination of the foot.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of chronic plantar fasciitis that have persisted for at least 6 months. despite previous conservative treatment, including corticosteroid injections, autologous PRP injections, physiotherapy, use of orthoses and NSAIDs,
* age ≥ 18 years,
* written consent to participate in the study

Exclusion Criteria:

* previous foot surgery,
* advanced diabetes impeding healing,
* significant obesity,
* contraindications to anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) AnkleHindfoot Scale | 3 months - 60 months after the treatment
  This comprehensive scale evaluates various aspects of foot health, including pain levels, functionality, and alignment, and is widely recognized for its reliability in orthopedic studies

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Piontek, MD PhD, Principal Investigator — tomasz.piontek@rehasport.pl

IPD SHARING:
Plan to Share IPD: No